CLINICAL TRIAL: NCT01938833
Title: A Phase I/II Study of Romidepsin in Combination With Abraxane in Patients With Metastatic Inflammatory Breast Cancer
Brief Title: Romidepsin and Abraxane in Treating Patients With Metastatic Inflammatory Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed by Sponsor
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13C.387; 2013-035 (Other: CCRRC); JT 2987 (Other: JeffTrial Number)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: HER2-negative Breast Cancer; Inflammatory Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms, Male; Breast Neoplasms | interventions — romidepsin; Depsipeptides; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Romidepsin and Abraxane) (Experimental): Patients receive abraxane IV over 30 minutes and romidepsin IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Romidepsin; Drug: Abraxane

INTERVENTIONS:
Drug: Romidepsin
  Other Names: Istodax; FK228; FR901228; Depsipeptide
Drug: Abraxane
  Other Names: Protein-bound paclitaxel; Paclitaxel albumin-stabilized nanoparticle formulation

SUMMARY:
This phase I/II trial studies the side effects and best dose of romidepsin when given together with paclitaxel albumin-stabilized nanoparticle formulation and to see how well they work in treating patients with metastatic inflammatory breast cancer. Romidepsin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving romidepsin and paclitaxel albumin-stabilized nanoparticle formulation may be an effective treatment for inflammatory breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To assess the safety of the combination of romidepsin plus Abraxane (paclitaxel albumin-stabilized nanoparticle formulation) delivered weekly. (Phase I)
2. To determine the maximum tolerated dose (MTD) of romidepsin with full dose weekly Abraxane to define a recommended phase II doses of the combination. (Phase I)
3. To assess the progression-free survival (PFS) in patients with human epidermal growth factor receptor 2 (HER2) negative, newly diagnosed metastatic inflammatory breast cancer treated with the combination of romidepsin and Abraxane. (Phase II)

SECONDARY OBJECTIVES:

1. To assess the safety and tolerability of the combination of romidepsin and Abraxane.
2. To determine the adverse event profile of the combination of romidepsin and Abraxane.
3. To assess the overall response rate (ORR) and clinical benefit rate (CBR) in patients with newly recurrent inflammatory breast cancer (IBC) treated with the combination of romidepsin and Abraxane.

OUTLINE: This is a phase I, dose-escalation study of romidepsin followed by a phase II study.

Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes and romidepsin IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed breast carcinoma with a clinical diagnosis of IBC based on the presence of inflammatory changes in the involved breast, such as diffuse erythema and edema (peau d'orange), with or without an underlying palpable mass involving the majority of the skin of the breast. Pathological evidence of dermal lymphatic invasion should be noted but is not required for diagnosis.
2. Patients may have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1 as described in detail in section 11.0 or non-measurable tumors
3. Patients must have demonstrated metastatic disease and not received >2 lines of systemic therapy for metastatic disease
4. Age > 18 years
5. ECOG performance status 0, 1 or 2
6. Patients must have normal organ and marrow function as defined below: a) Leukocytes > 2,500/mcL b) Absolute neutrophil count > 1,500/mcL c) Hemoglobin > 9 g/dl d) Platelets > 100,000/mcL e) Total bilirubin < 1.5 mg/dl f) AST/ALT (SGOT/SGPT) < 2.5 x ULN g) Alkaline Phosphatase < 2.5 x ULN (unless bone metastasis is present in the absence of liver metastasis, in which case 3.0 x ULN would be acceptable. h) Serum magnesium > 1.8 mg/dL i) Serum creatinine < 1.5 mg/dl j) Serum potassium > 3.8 mmol/L
7. Tumor negative for HER2 expression (0 or 1+ by IHC) or negative FISH testing
8. Patients must have a life expectancy of at least 12 weeks
9. Patients must be recovered from the effects of any prior surgery, radiotherapy, or other antineoplastic therapy
10. Patients must have < Grade 2 pre-existing peripheral neuropathy per CTCAE
11. Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment
12. Negative serum or urine β-hCG pregnancy test at screening, performed no more than 72 hours prior to treatment initiation; for patients of childbearing potential
13. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse event from agents administered more than 4 weeks earlier
2. Patients may not be receiving any other investigational agents or active anti-neoplastic therapies
3. Patients who have previously received romidepsin or Abraxane
4. Patients with untreated or uncontrolled brain metastases or leptomeningeal disease
5. Patients with known hypersensitivity to any of the components of romidepsin or who have had hypersensitivity reactions to paclitaxel
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
7. Any known cardiac abnormalities such as:

   1. Congenital long QT syndrome
   2. QTc interval ≥ 500 milliseconds
   3. Myocardial infarction within 6 months of C1D1. Subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate
   4. Other significant EKG abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min)
   5. Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV (see Appendix III) In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
   6. An EKG recorded at screening showing evidence of cardiac ischemia (ST depression depression of ≥2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present
   7. Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions (see Appendix IV) and/or known ejection fraction <40% by MUGA or <50% by echocardiogram and/orMRI
   8. A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD)
   9. Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes
   10. Uncontrolled hypertension, i.e., blood pressure (BP) of ≥ 160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria
   11. Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
   12. Patients taking drugs leading to significant QT prolongation (See Appendix I: Medications That May Cause QTc Prolongation)
   13. Concomitant use of CYP3A4 inhibitors (see Appendix II)
8. Patients with known HIV, hepatitis B or C (However, if patients have previously been treated for hepatitis B or C and have undetectable viral loads, they can be considered eligible for trial)
9. Pregnant or breast feeding. Refer to section 4.4 for further detail
10. Patients with any other medical or psychological condition deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-khalaf, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Blum JL, Savin MA, Edelman G, Pippen JE, Robert NJ, Geister BV, Kirby RL, Clawson A, O'Shaughnessy JA. Phase II study of weekly albumin-bound paclitaxel for patients with metastatic breast cancer heavily pretreated with taxanes. Clin Breast Cancer. 2007 Dec;7(11):850-6. doi: 10.3816/CBC.2007.n.049. PMID 18269774
- [Background] Chang H, Jeung HC, Jung JJ, Kim TS, Rha SY, Chung HC. Identification of genes associated with chemosensitivity to SAHA/taxane combination treatment in taxane-resistant breast cancer cells. Breast Cancer Res Treat. 2011 Jan;125(1):55-63. doi: 10.1007/s10549-010-0825-z. Epub 2010 Mar 12. PMID 20224928
- [Background] Chang H, Rha SY, Jeung HC, Jung JJ, Kim TS, Kwon HJ, Kim BS, Chung HC. Identification of genes related to a synergistic effect of taxane and suberoylanilide hydroxamic acid combination treatment in gastric cancer cells. J Cancer Res Clin Oncol. 2010 Dec;136(12):1901-13. doi: 10.1007/s00432-010-0849-0. Epub 2010 Mar 9. PMID 20217129
- [Background] Chang S, Parker SL, Pham T, Buzdar AU, Hursting SD. Inflammatory breast carcinoma incidence and survival: the surveillance, epidemiology, and end results program of the National Cancer Institute, 1975-1992. Cancer. 1998 Jun 15;82(12):2366-72. PMID 9635529
- [Background] Chen MY, Liao WS, Lu Z, Bornmann WG, Hennessey V, Washington MN, Rosner GL, Yu Y, Ahmed AA, Bast RC Jr. Decitabine and suberoylanilide hydroxamic acid (SAHA) inhibit growth of ovarian cancer cell lines and xenografts while inducing expression of imprinted tumor suppressor genes, apoptosis, G2/M arrest, and autophagy. Cancer. 2011 Oct 1;117(19):4424-38. doi: 10.1002/cncr.26073. PMID 21491416
- [Background] Cristofanilli M, Buzdar AU, Hortobagyi GN. Update on the management of inflammatory breast cancer. Oncologist. 2003;8(2):141-8. doi: 10.1634/theoncologist.8-2-141. PMID 12697939
- [Background] Colpaert CG, Vermeulen PB, Benoy I, Soubry A, van Roy F, van Beest P, Goovaerts G, Dirix LY, van Dam P, Fox SB, Harris AL, van Marck EA. Inflammatory breast cancer shows angiogenesis with high endothelial proliferation rate and strong E-cadherin expression. Br J Cancer. 2003 Mar 10;88(5):718-25. doi: 10.1038/sj.bjc.6600807. PMID 12618881
- [Background] Desai N, Trieu V, Yao R, et al. Increased transport of nanoparticle albumin-bound paclitaxel (ABI-007) by endothelial gp60-mediated caveolar transcytosis: a pathway inhibited by Taxol. Eur J Cancer Suppl. 2004;2:182.
- [Background] Gradishar WJ, Krasnojon D, Cheporov S, Makhson AN, Manikhas GM, Clawson A, Bhar P. Significantly longer progression-free survival with nab-paclitaxel compared with docetaxel as first-line therapy for metastatic breast cancer. J Clin Oncol. 2009 Aug 1;27(22):3611-9. doi: 10.1200/JCO.2008.18.5397. Epub 2009 May 26. PMID 19470941
- [Background] Kim H, Kim SN, Park YS, Kim NH, Han JW, Lee HY, Kim YK. HDAC inhibitors downregulate MRP2 expression in multidrug resistant cancer cells: implication for chemosensitization. Int J Oncol. 2011 Mar;38(3):807-12. doi: 10.3892/ijo.2010.879. Epub 2010 Dec 17. PMID 21170509
- [Background] Hoshino I, Matsubara H, Akutsu Y, Nishimori T, Yoneyama Y, Murakami K, Komatsu A, Sakata H, Matsushita K, Ochiai T. Gene expression profiling induced by histone deacetylase inhibitor, FK228, in human esophageal squamous cancer cells. Oncol Rep. 2007 Sep;18(3):585-92. PMID 17671705
- [Background] Lassen U, Molife LR, Sorensen M, Engelholm SA, Vidal L, Sinha R, Penson RT, Buhl-Jensen P, Crowley E, Tjornelund J, Knoblauch P, de Bono JS. A phase I study of the safety and pharmacokinetics of the histone deacetylase inhibitor belinostat administered in combination with carboplatin and/or paclitaxel in patients with solid tumours. Br J Cancer. 2010 Jun 29;103(1):12-7. doi: 10.1038/sj.bjc.6605726. Epub 2010 Jun 15. PMID 20588278
- [Background] Low JA, Berman AW, Steinberg SM, Danforth DN, Lippman ME, Swain SM. Long-term follow-up for locally advanced and inflammatory breast cancer patients treated with multimodality therapy. J Clin Oncol. 2004 Oct 15;22(20):4067-74. doi: 10.1200/JCO.2004.04.068. PMID 15483018
- [Background] Modesitt SC, Sill M, Hoffman JS, Bender DP; Gynecologic Oncology Group. A phase II study of vorinostat in the treatment of persistent or recurrent epithelial ovarian or primary peritoneal carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2008 May;109(2):182-6. doi: 10.1016/j.ygyno.2008.01.009. Epub 2008 Mar 4. PMID 18295319
- [Background] Nguyen DM, Sam K, Tsimelzon A, Li X, Wong H, Mohsin S, Clark GM, Hilsenbeck SG, Elledge RM, Allred DC, O'Connell P, Chang JC. Molecular heterogeneity of inflammatory breast cancer: a hyperproliferative phenotype. Clin Cancer Res. 2006 Sep 1;12(17):5047-54. doi: 10.1158/1078-0432.CCR-05-2248. PMID 16951220
- [Background] Nyman DW, Campbell KJ, Hersh E, Long K, Richardson K, Trieu V, Desai N, Hawkins MJ, Von Hoff DD. Phase I and pharmacokinetics trial of ABI-007, a novel nanoparticle formulation of paclitaxel in patients with advanced nonhematologic malignancies. J Clin Oncol. 2005 Nov 1;23(31):7785-93. doi: 10.1200/JCO.2004.00.6148. PMID 16258082
- [Background] Rasheed W, Bishton M, Johnstone RW, Prince HM. Histone deacetylase inhibitors in lymphoma and solid malignancies. Expert Rev Anticancer Ther. 2008 Mar;8(3):413-32. doi: 10.1586/14737140.8.3.413. PMID 18366289
- [Background] Robertson FM, Woodward WA, Pickei R, Ye Z, Bornmann W, Pal A, Peng Z, Hall CS, Cristofanilli M. Suberoylanilide hydroxamic acid blocks self-renewal and homotypic aggregation of inflammatory breast cancer spheroids. Cancer. 2010 Jun 1;116(11 Suppl):2760-7. doi: 10.1002/cncr.25176. PMID 20503408
- [Background] Sasakawa Y, Naoe Y, Sogo N, Inoue T, Sasakawa T, Matsuo M, Manda T, Mutoh S. Marker genes to predict sensitivity to FK228, a histone deacetylase inhibitor. Biochem Pharmacol. 2005 Feb 15;69(4):603-16. doi: 10.1016/j.bcp.2004.11.008. Epub 2004 Dec 23. PMID 15670579
- [Background] ten Tije AJ, Verweij J, Loos WJ, Sparreboom A. Pharmacological effects of formulation vehicles : implications for cancer chemotherapy. Clin Pharmacokinet. 2003;42(7):665-85. doi: 10.2165/00003088-200342070-00005. PMID 12844327
- [Background] Ueda H, Nakajima H, Hori Y, Goto T, Okuhara M. Action of FR901228, a novel antitumor bicyclic depsipeptide produced by Chromobacterium violaceum no. 968, on Ha-ras transformed NIH3T3 cells. Biosci Biotechnol Biochem. 1994 Sep;58(9):1579-83. doi: 10.1271/bbb.58.1579. PMID 7765477
- [Background] Van Laere S, Van der Auwera I, Van den Eynden GG, Fox SB, Bianchi F, Harris AL, van Dam P, Van Marck EA, Vermeulen PB, Dirix LY. Distinct molecular signature of inflammatory breast cancer by cDNA microarray analysis. Breast Cancer Res Treat. 2005 Oct;93(3):237-46. doi: 10.1007/s10549-005-5157-z. PMID 16172796
- [Background] Zou CF, Jia L, Jin H, Yao M, Zhao N, Huan J, Lu Z, Bast RC Jr, Feng Y, Yu Y. Re-expression of ARHI (DIRAS3) induces autophagy in breast cancer cells and enhances the inhibitory effect of paclitaxel. BMC Cancer. 2011 Jan 19;11:22. doi: 10.1186/1471-2407-11-22. PMID 21244707
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Romidepsin and Abraxane): Patients receive abraxane IV over 30 minutes and romidepsin IV over 60 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Romidepsin
  Abraxane
Period: Overall Study
Arm/Group | Treatment (Romidepsin and Abraxane)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Romidepsin and Abraxane)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum-Tolerated Dose of Romidepsin (Phase I)
Description: Determined according to incidence of dose-limiting toxicity, graded using the National Cancer Institute (NCI) CTCAE version 4.0
Time Frame: 28 days
Population: Data were not collected and the Outcome will never be analyzed.
Arm/Group | Treatment (Romidepsin and Abraxane)
Number analyzed (Participants) | 0

2. Primary Outcome: Progression-Free Survival (PFS)
Time Frame: The duration of time from start of treatment to time of progression or death, whichever occurs first, assessed up to 5 years
Population: Data were not collected and the Outcome will never be analyzed
Arm/Group | Treatment (Romidepsin and Abraxane)
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Adverse Events, Graded According to NCI CTCAE Version 4.0
Description: Summary tables of grade 2, 3, and 4 toxicities, adverse events (AE), and serious adverse events (SAE) will be generated at the conclusion of the study as well as at the conclusion of phase I study and after 15 patients have been collected on at the interim evaluation time point of the phase 2 part of the study.
Time Frame: Up to 30 days
Population: Data were not collected and the Outcome will never be analyzed.
Arm/Group | Treatment (Romidepsin and Abraxane)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Rate (ORR)
Description: The 95% confidence intervals should be provided.
Time Frame: Up to 5 years
Population: Data were not collected and the Outcome will never be analyzed.
Arm/Group | Treatment (Romidepsin and Abraxane)
Number analyzed (Participants) | 0

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The 95% confidence intervals should be provided.
Time Frame: Up to 5 years
Population: Data were not collected and the Outcome will never be analyzed.
Arm/Group | Treatment (Romidepsin and Abraxane)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Romidepsin and Abraxane)
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Romidepsin and Abraxane) (N=7)
Catheter related Infection (Renal and urinary disorders) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Romidepsin and Abraxane) (N=9)
Alanine Aminotransferase Increased (Blood and lymphatic system disorders) | 3 (10)
Alkaline phosphatase Increased (Blood and lymphatic system disorders) | 2 (2)
Alopecia (Immune system disorders) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 7 (18)
Anorexia (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate Aminotransferase increased (Blood and lymphatic system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (2)
Body Aches (General disorders) | 1 (1)
Bone Pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (General disorders) | 4 (4)
Dry mouth (General disorders) | 1 (1)
Dsygeusia (General disorders) | 3 (4)
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Edema in the Limbs (General disorders) | 4 (9)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Eye disorders (Eye disorders) | 2 (4)
Fatigue (General disorders) | 5 (11)
Fever (Infections and infestations) | 1 (1)
Flu like symptoms-Cold (Infections and infestations) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Gastrointestinal other symptoms (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1)
Headaches (General disorders) | 5 (5)
Heart Burn (Gastrointestinal disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 6 (14)
Hyperphosphatemia (Blood and lymphatic system disorders) | 1 (2)
Hypocalcemia (Blood and lymphatic system disorders) | 2 (2)
Hypokalemia (Blood and lymphatic system disorders) | 1 (2)
Hyponatremia (Blood and lymphatic system disorders) | 2 (4)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (2)
INR increased (Blood and lymphatic system disorders) | 1 (2)
Insomnia (Nervous system disorders) | 2 (2)
Interstitial Cystitis (Renal and urinary disorders) | 1 (1)
Irregular Menstruation (Reproductive system and breast disorders) | 1 (1)
LDH increased (Endocrine disorders) | 1 (1)
Lower Back Spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower Jaw Infection (Infections and infestations) | 1 (1)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 1 (6)
Malaise (General disorders) | 1 (1)
Mucositis oral (General disorders) | 1 (1)
Lump (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6)
Neuropathy (Nervous system disorders) | 4 (7)
Neutrophil count decreased (Infections and infestations) | 4 (7)
Numbness (Nervous system disorders) | 1 (1)
Pain (General disorders) | 7 (17)
Platelet Count decreased (Blood and lymphatic system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Negative Thoughts (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Right Foot Pain (General disorders) | 1 (1)
Right leg pain (General disorders) | 1 (1)
Runny Nose (General disorders) | 1 (1)
Sensory Neuropathy (Nervous system disorders) | 2 (2)
Shoulder pain (General disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin Disorder - Hole (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Infection-Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Peeling (Skin and subcutaneous tissue disorders) | 1 (1)
Sore Throat (General disorders) | 1 (1)
Tightness (Musculoskeletal and connective tissue disorders) | 2 (9)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Toothache (General disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (1)
Urine Culture Growth (Renal and urinary disorders) | 1 (2)
Vaginal Dryness (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
White blood cell decreased (Infections and infestations) | 5 (12)
Wound - Right Arm (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes